CLINICAL TRIAL: NCT00229112
Title: A Prospective, Multicenter, Double-Blind With In-House Blinding, Randomized, Comparative Study to Evaluate the Efficacy, Safety, and Tolerability, of Ertapenem Versus Piperacillin/Tazobactam in the Treatment of Diabetic Foot Infections in Adults.
Brief Title: Comparative Study of Ertapenem Versus Another Antibiotic in the Treatment of Diabetic Foot Infections in Adults (0826-034)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0826-034; 2005_083
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Foot Infections in Diabetic Patients
MeSH Terms: interventions — Ertapenem; Duration of Therapy; Tazobactam

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0826, ertapenem sodium / Duration of Treatment - 24 weeks
Drug: Comparator: Piperacillin/Tazobactam / Duration of Treatment - 24 weeks

SUMMARY:
This study will compare the efficacy, safety and tolerability of intravenous ertapenem versus another intravenous antibiotic in the treatment of moderate to severe diabetic foot infections.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 Diabetes Mellitus treated with diet or medication
* Clinically or microbiologically documented foot infection below the knee
* Osteomyelitic bone must be removed within 48 hours of study entry

Exclusion Criteria:

* Uncomplicated skin infections
* Infected burn wounds
* Necrotizing fascitis
* Wounds with gangrene that cannot be removed with debridement
* Infections of prosthetic materials
* Foreign materials that can not be removed by surgical debridement
* Patients with another antibiotic 3 days prior to enrollment without evidence of treatment failure and presence of a positive culture
* Insufficient blood flow to the limb requiring a revascularization procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2001-04; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Clinical Cure/Improvement at discontinuation of IV antibiotic therapy.

SECONDARY OUTCOMES:
Clinical Cure: 1. Day 5 of IV antibiotic therapy; 2.10 days after completion of all antibiotic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Citron DM, Goldstein EJ, Merriam CV, Lipsky BA, Abramson MA. Bacteriology of moderate-to-severe diabetic foot infections and in vitro activity of antimicrobial agents. J Clin Microbiol. 2007 Sep;45(9):2819-28. doi: 10.1128/JCM.00551-07. Epub 2007 Jul 3. PMID 17609322
- [Background] Armstrong DG, Lipsky BA, Polis AB, Abramson MA. Does dermal thermometry predict clinical outcome in diabetic foot infection? Analysis of data from the SIDESTEP* trial. Int Wound J. 2006 Dec;3(4):302-7. doi: 10.1111/j.1742-481X.2006.00269.x. PMID 17199766
- [Background] Lipsky BA, Sheehan P, Armstrong DG, Tice AD, Polis AB, Abramson MA. Clinical predictors of treatment failure for diabetic foot infections: data from a prospective trial. Int Wound J. 2007 Mar;4(1):30-8. doi: 10.1111/j.1742-481X.2006.00274.x. PMID 17425547
- [Background] Lipsky BA, Polis AB, Lantz KC, Norquist JM, Abramson MA. The value of a wound score for diabetic foot infections in predicting treatment outcome: a prospective analysis from the SIDESTEP trial. Wound Repair Regen. 2009 Sep-Oct;17(5):671-7. doi: 10.1111/j.1524-475X.2009.00521.x. Epub 2009 Aug 11. PMID 19671126
- [Result] Lipsky BA, Armstrong DG, Citron DM, Tice AD, Morgenstern DE, Abramson MA. Ertapenem versus piperacillin/tazobactam for diabetic foot infections (SIDESTEP): prospective, randomised, controlled, double-blinded, multicentre trial. Lancet. 2005 Nov 12;366(9498):1695-703. doi: 10.1016/S0140-6736(05)67694-5. PMID 16291062
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html